CLINICAL TRIAL: NCT02282254
Title: An Open-label, Randomized, Cross-over Study to Assess the Efficacy of Single-hormone and Dual-hormone Closed-loop Strategy in Regulating Overnight Glucose Levels in Type 1 diabètes Adults With Hypoglycemia Unawareness and Documented Nocturnal Hypoglycemia
Brief Title: Closed-loop Control of Overnight Glucose Levels (Artificial Pancreas) in Type 1 Diabètes Adults With Hypoglycemia Unawareness and Documented Nocturnal Hypoglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-09
Record Dates: First submitted 2014-10-19; First posted 2014-11-04 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia unawareness; Nocturnal hypoglycemia; Closed-loop strategy; Artificial pancreas; Glucagon; Hypoglycemia; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-hormone closed-loop strategy (Active Comparator)
  Interventions: Other: Overnight intervention
- Dual-hormone closed-loop strategy (Active Comparator)
  Interventions: Other: Overnight intervention

INTERVENTIONS:
Other: Overnight intervention — Subjects will be admitted at the research facility at 19:00. A cannula will be inserted into an arm or a hand vein for blood sampling purposes. On dual-hormone closed-loop visits, glucagon will be reconstituted according to the manufacturer's instructions and a MiniMed® Paradigm® Veo™ pump containing the glucagon solution will be installed. At 20:30, a snack containing 20g of carbohydrate will be given. Closed-loop strategy will start at 20:00 until 7:00 next morning. A glucose sensor reading will be entered manually in a tablet every 10 minutes. The tablet will generate a recommendation for the basal rates of insulin delivery and glucagon mini-boluses (glucagon recommendations will only be generated during the dual hormone closed-loop visits). Pumps' parameters will then be changed manually to implement the tablet generated recommendations.

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop strategy would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

The main objective of this project is to compare the efficacy of single-hormone and dual-hormone closed-loop strategy to regulate overnight glucose levels in a in-patient study in type 1 diabetes adults with hypoglycemia unawareness and documented nocturnal hypoglycemia.

The investigators hypothesized that dual-hormone closed-loop strategy is more effective in regulating overnight glucose levels compared to single-hormone closed-loop strategy.

DETAILED DESCRIPTION:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop strategy would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

The investigators aim to conduct the 1st randomized cross-over trial comparing single- hormone and dual-hormone closed-loop strategy to regulate overnight glucose levels. The investigators aim to compare the two interventions for 10 hours in two subgroups of adults with type 1 diabètes. Patients from both subgroups will present documented nocturnal hypoglycemia. One subgroup will consist of patients with hypoglycemia unawareness while the other subgroup will consist of patients with hypoglycemia unawareness. This study will allow to determine if there is a greater benefit of a closed-loop strategy in a higher-risk hypoglycemia unaware group.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. HbA1c ≤ 12%.
5. Hypoglycemia awareness or unawareness assessed by a questionnaire.
6. Documented NH during the run-in period.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Pregnancy.
4. Severe hypoglycemic episode within two weeks of screening.
5. Current use of glucocorticoid medication (except low stable dose).
6. Known or suspected allergy to the trial products or snack contents.
7. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
8. Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport).
9. Failure to comply with team's recommendations (e.g. not willing to eat snacks, not willing to change pump parameters, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose levels spent below 4 mmol/L | Up to 8 hours

SECONDARY OUTCOMES:
Percentage of time of plasma glucose levels spent between 4 and 8 mmol/L | Up to 8 hours
Percentage of time of plasma glucose levels spent between 4 and 10 mmol/L | Up to 8 hours
Percentage of time of plasma glucose levels spent below 3.5 mmol/L | Up to 8 hours
Percentage of time of plasma glucose levels spent below 3.3. mmol/L | Up to 8 hours
Percentage of time of plasma glucose levels spent above 8 mmol/L | Up to 8 hours
Percentage of time of plasma glucose levels spent above 10 mmol/L | Up to 8 hours
Area under the curve of plasma glucose levels spent below 4 mmol/L | Up to 8 hours
Area under the curve of plasma glucose levels spent below 3.5 mmol/L | Up to 8 hours
Area under the curve of plasma glucose levels spent below 3.3 mmol/L | Up to 8 hours
Area under the curve of plasma glucose levels spent above 8 mmol/L | Up to 8 hours
Area under the curve of plasma glucose levels spent above 10 mmol/L | Up to 8 hours
Mean plasma glucose levels | Up to 8 hours
Standard deviation of plasma glucose levels | Up to 8 hours
Total insulin delivery | Up to 8 hours
Total glucagon delivery | Up to 8 hours
Number of subjects experiencing at least one hypoglycemic event requiring oral treatment | Up to 8 hours
Total number of hypoglycemic events requiring treatment | Up to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Abitbol A, Rabasa-Lhoret R, Messier V, Legault L, Smaoui M, Cohen N, Haidar A. Overnight Glucose Control with Dual- and Single-Hormone Artificial Pancreas in Type 1 Diabetes with Hypoglycemia Unawareness: A Randomized Controlled Trial. Diabetes Technol Ther. 2018 Mar;20(3):189-196. doi: 10.1089/dia.2017.0353. Epub 2018 Feb 2. PMID 29393675